CLINICAL TRIAL: NCT06492889
Title: Randomized Trial Comparing Progestin With Mifepristone Versus Mifepristone Alone for Use as Missed Period Pills
Brief Title: Assessing the Efficacy and Acceptability of Two Missed Period Pills Regimens
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Cuidado Integral de la Mujer, Gineclinic, S.C. (Unknown); Servicios de Salud Medieg, A. C (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8007
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy Early; Pregnancy Related
MeSH Terms: interventions — Levonorgestrel; Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levonorgestrel plus mifepristone (Experimental): Women randomized to take one pill containing 1.5 mg levonorgestrel followed one to two days later by 200 mg mifepristone.
  Interventions: Drug: Levonorgestrel; Drug: Mifepristone
- Placebo plus mifepristone (Experimental): Women randomized to take one placebo pill followed one to two days later by 200 mg mifepristone.
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Levonorgestrel — Participants in the levonorgestrel plus mifepristone group will receive one tablet of 1.5 mg levonorgestrel
  Arms: Levonorgestrel plus mifepristone
Drug: Mifepristone — Participants in both groups will receive one tablet of 200 mg mifepristone

SUMMARY:
The goal of this trial is to examine the efficacy and acceptability of two medication regimens at inducing a return of menses when used 2-8 days after a missed period. The first regimen consists of one dose of 1.5 mg levonorgestrel followed one to two days later by one dose of 200 mg mifepristone. The second regimen will consist of one dose of a placebo pill, followed one to two days later by one dose of 200 mg mifepristone.

The investigators will assess and compare the efficacy of both regimens (proportion of women in each group not pregnant at follow-up who were determined to be pregnant at enrollment), and the effectiveness of both regimens (proportion of all participants not pregnant at follow-up among all participants enrolled)

ELIGIBILITY:
Inclusion Criteria:

* Age 15-49 years
* General good health
* Does not want to be pregnant
* History of regular monthly menstrual cycles (+/- 3 days)
* Missed menses of 2 to 8 days
* Sexual activity in the past month
* Willing and able to sign consent forms
* Willing to return for a follow-up visit
* Willing to provide urine sample at enrollment and follow-up

Exclusion Criteria:

* Known allergies or contraindications to either study drug
* Symptoms or risk factors for ectopic pregnancy
* Current use of an IUD, contraceptive implant or injectable

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 286 (Estimated)
Dates: Start 2024-07-22 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the missed period pills regimen | Two weeks
  Proportion of women not pregnant at follow-up who were determined to be pregnant at enrollment
Effectiveness of the missed period pills regimen | Two weeks
  Proportion of women not pregnant at follow-up among all women enrolled, including those who were pregnant and not pregnant at enrollment

SECONDARY OUTCOMES:
Effectiveness at inducing return of menses within 10 days of missed menses | One to two weeks
  Proportion of participants who experience menstrual bleeding after taking the study medications
Safety/side effects | Two weeks
  Incidence of side effects and complications
Acceptability | Two weeks
  Proportion of participants who report that the missed period pills service was acceptable or highly acceptable

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects